CLINICAL TRIAL: NCT07022925
Title: An Observational Virtual Trial to Investigate the Accuracy of a Wearable Device in Collecting Data Related to Perimenopausal Symptoms in Women
Brief Title: A Trial to Investigate the Accuracy of a Wearable Device in Collecting Data Related to Perimenopausal Symptoms in Women
Status: Recruiting | Type: Observational
Sponsor: IdentifyHer Limited (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 24IDCFI01
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Perimenopause; Perimenopausal Depression; Perimenopausal Insomnia; Perimenopausal Women; Menopausal Depression; Menopausal Hot Flashes; Menopausal and Postmenopausal Disorders; Menopausal Vasomotor Symptoms
Keywords: Menopause; Perimenopause; Vasomotor symptoms; Hot flashes; IdentifyHer; Peri; Perimenopausal symptoms
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IndentifyHer's Peri: IndentifyHer's Peri investigational device is a commercial, non-invasive, wearable sensor that works in combination with a digital platform to quantify and profile the frequency and severity of perimenopausal symptoms including hot flashes, night sweats, anxiety, and sleep disturbances.

SUMMARY:
The goal of this observational study is to investigate the accuracy of the device in characterizing perimenopausal and menopausal symptoms including vasomotor symptoms, anxiety, sleep quality compared to self-reported symptoms via an app. The main question it aims to answer is:

What is the accuracy of the developed algorithm from the investigational device compared to daily self-report via an app in characterizing perimenopausal symptoms?

Participants will be asked to wear IndentifyHer's wearable non-invasive sensor and complete a daily electronic diary and questionnaires on stress, anxiety, and sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Females between 35-55 years of age, inclusive
2. Self-reported perimenopausal women experiencing hot flushes or night sweats
3. Individuals of child-bearing potential must confirm they are not pregnant, do not plan to become pregnant, and agree to use a medically approved method of birth control for the duration of the study. Acceptable methods of birth control include:

   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence
4. Agrees to maintain current lifestyle as much as possible throughout the study, including diet, exercise, supplements/medications, and sleep
5. Provided voluntary and informed consent to participate in the study
6. Generally healthy as determined by medical history with no unstable diagnosed medical conditions

Exclusion Criteria:

1. Allergy or sensitivity to adhesive used for wearing the investigational device
2. Self-reported use of a pacemaker
3. Self-reported unstable diagnosed anxiety disorder
4. Self-reported sleep disorder requiring medical treatment
5. Self-reported skin conditions or sensitive skin around the area of application
6. Self-reported surgery in the past three months or individuals who have planned surgery during the course of the study
7. Alcohol intake average of ˃1 standard drink per day
8. Alcohol or drug abuse within the last 12 months that has required treatment
9. Current use of prescribed and/or over-the-counter (OTC) medications/supplements that may impact data recorded by the investigational device (see Section 7.3)
10. Participation in other clinical research studies 30 days prior to screening
11. Individuals who are unable to give informed consent
12. Any other condition or lifestyle factor, that may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: N/A - virtual study. Participants are recruited online.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing Vasomotor symptoms. | Day 0 to 14
  The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing vasomotor symptoms. Questionnaire answers include "not at all" to "extremely".
The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing anxiety | Day 0 to 14
  The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing anxiety. Questionnaire answers include "not at all" to "nearly everyday".
The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing sleep quality | Day 0 to 14
  The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing sleep quality. Questionnaire answers include "terrible" to "very well".
The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing perimenopausal symptoms considering confounders | Day 0 to 14
  The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing perimenopausal symptoms considering confounders of warmer environmental conditions. Questionnaire answers include "not at all" to "nearly all day".
The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing perimenopausal symptoms considering confounders | Day 0 to 14
  The accuracy of the developed algorithm from the investigational device compared to daily self-report questionnaire via an app in characterizing perimenopausal symptoms considering confounders of an ethnically-diverse study population. Questionnaire answers include "not at all" to "nearly all day".

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada